CLINICAL TRIAL: NCT01867827
Title: Real-time fMRI Neurofeedback for Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Principal Investigator, David Linden, Professor of Translational Neuroscience, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPON997-11
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Neurofeedback; Exercise

ARMS (2):
- Neurofeedback and Physical Exercise (Experimental): This group will undergo neurofeedback intervention in the fMRI scanner in weeks 1,5 and 12. They will also undergo physical exercise training on WiiFit device once a week after the first month till the end of the study at 12 weeks.
  Interventions: Other: Neurofeedback and Physical Exercise
- Physical Exercise (Active Comparator): This group will undergo Physical Exercise intervention on the WiiFit device 3 times a week in the first month and once a week after the first month till the end of the study at 12 weeks.
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Neurofeedback and Physical Exercise
  Arms: Neurofeedback and Physical Exercise
Other: Physical Exercise
  Arms: Physical Exercise

SUMMARY:
The aim of the study is to train patients with Parkinson's Disease to increase activity in a brain area that is involved in the control of motor functions with the use of a technique called real-time fMRI neurofeedback (NF) along with regular physical exercise. This will be a randomised and controlled clinical trial to evaluate the benefits of a novel treatment. The investigators expect NF training along with physical exercise practise to better improve motor functions compared to physical exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* People with Parkinson's Disease
* Hoehn and Yahr stages 1-3 of the disease

Exclusion Criteria:

* Patients with dementia or significant comorbidity
* those who fail the safety screening to go into an MRI scanner
* those who cannot travel to the University

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the 'Movement Disorder Society - Unified Parkinson's Disease Rating Scale' (MDS-UPDRS) | Change from Baseline in the 'Movement Disorder Society - Unified Parkinson's Disease Rating Scale' (MDS-UPDRS) in 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the 'Parkinson's Disease Questionnaire 39' (PDQ-39) | Change from baseline in the 'Parkinson's Disease Questionnaire 39' (PDQ-39) at 4 weeks
Change from baseline in the 'Parkinson's Disease Questionnaire 39' (PDQ-39) | Change from baseline in the 'Parkinson's Disease Questionnaire 39' (PDQ-39) in 12 weeks
Change from baseline in the 'Actigraph' | Change from baseline in the 'Actigraph' at 12 weeks
Change from baseline in the 'GaitRite' | Change from baseline in the 'GaitRite' at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Linden, MD, PhD, Principal Investigator — Cardiff University
Locations (1):
- School of Medicine, Cardiff University, Cardiff, Wales, United Kingdom

REFERENCES:
- See also: Paper reporting trial results — https://doi.org/10.3389/fnbeh.2016.00111